CLINICAL TRIAL: NCT07375134
Title: Evaluation of the Relationship Between Flexor Retinacular Ligament Thickness and the Development of Heel Pain Syndrome After Carpal Tunnel Surgery.
Brief Title: Observational Study - Heel Syndrome and Relationship to Flexor Retinacular Ligament Thickness
Acronym: ESTEREL
Status: Active, not recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: COS-RGDS-2023-12-034-P-DINH-A
Record Dates: First submitted 2025-11-25; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome (CTS); Heel Pain Syndrome
Keywords: heel pain syndrome; patients operated on for carpal tunnel syndrome; thickness of the flexor retinacular ligament
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with heel-of-hand syndrome 6 months after surgery for carpal tunnel syndrome: Patients with heel of the hand syndrome, 6 months after surgery for carpal tunnel syndrome (measurement of retinacular ligament thickness intraoperatively)
- Patients without heel of the hand syndrome 6 months after surgery for carpal tunnel syndrome: Patients without heel of the hand syndrome, 6 months after surgery for carpal tunnel syndrome (measurement of retinacular ligament thickness intraoperatively)

SUMMARY:
Numerous studies have examined the relationship between carpal tunnel syndrome and the thickness of the flexor retinacular ligament. This varies along the course of the median nerve (the distal portion being the thickest) and increases with age. These studies have shown that the thickness of the ligament is greater in patients with carpal tunnel syndrome, without, however, demonstrating that it is related to the onset of this syndrome. According to Bartolomé-Villar, it may rather influence the onset of carpal pain.

The objective of this study is to determine whether a relationship exists between the thickness of the flexor retinacular ligament and the development of heel syndrome in the postoperative period for carpal tunnel syndrome.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, single-center, open-label observational study conducted on a population of patients operated on for carpal tunnel syndrome.

This study does not alter patient care or the doctor-patient relationship. Evaluations take place during routinely scheduled consultations. The frequency of evaluations is consistent with standard postoperative follow-up.

ELIGIBILITY:
Inclusion Criteria :

* Male or female patient over 18 years of age
* Patient who has been informed of the research and has not indicated their opposition to the use of their medical data
* Patient who is a candidate for first-time carpal tunnel surgery

Exclusion Criteria :

* Emergency surgery performed in a post-traumatic context
* Mental impairment or any other reason that may hinder understanding or strict application of the protocol
* Patient not affiliated with the French social security system
* Patient under legal protection, guardianship, or curatorship
* Patient already included in another therapeutic study protocol

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated on for carpal tunnel syndrome by the same operator using the Chow technique.
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Compare the intraoperative measurement of flexor retinacular ligament thickness between the two groups of patients operated on for carpal tunnel syndrome by the same surgeon using the Chow technique (with and without hand heel syndrome). | perioperatively
  Intraoperative measurement of flexor retinacular ligament thickness

SECONDARY OUTCOMES:
Assess the existence of other factors that may be related to the occurrence of hand heel syndrome (Spontaneous pain) according to the initial characteristics and follow-up data of patients with and without hand heel syndrome. | Baseline to six months after the surgery
  Spontaneous pain in the heel of the hand assessed by the patient on a simple numeric rating scale (SNS) from 0 to 10 (0 = no pain, 10 = maximum pain).
Assess the existence of other factors that may be linked to the occurrence of heel hand syndrome (Pain on palpation of the heel of the hand) based on initial characteristics and follow-up data, patients with and without hand heel syndrome | Baseline to six months after the surgery
  Pain on palpation of the heel of the hand assessed by the patient on a simple numeric rating scale (SNS) from 0 to 10 (0 = no pain, 10 = maximum pain).
Assess the existence of other factors that may be linked to the occurrence of heel hand syndrome (Postoperative complications) based on follow-up data, patients with and without hand heel syndrome | Immediately after the intervention to six months postoperatory
  Postoperative complications (inflammatory scar or keloid, complex regional pain syndrome, infection or hematoma).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio DINH, Dr, Principal Investigator — Hôpital Privé Paul d'Egine
Locations (1):
- Hôpital Privé Paul d'Egine, Champigny-sur-Marne, France